CLINICAL TRIAL: NCT01471574
Title: A Phase 3, Open Label Study of Safety and Efficacy With BMS-790052 Plus Peg-Interferon Alfa 2a and Ribavirin in Previously Untreated HCV Patients Coinfected With Human Immunodeficiency Virus (HIV) and Hepatitis C Virus (HCV)
Brief Title: Safety and Efficacy Study of Daclatasvir (BMS-790052) Plus Pegylated Interferon-Alfa 2a and Ribavirin in Patients Coinfected With Untreated Hepatitis C Virus and HIV Virus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI444-043; 2011-003067-30 (EudraCT Number)
Record Dates: First submitted 2011-11-04; First posted 2011-11-15 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2015-12

CONDITIONS: Hepatitis C, Genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Daclatsvir + Ribavirin + PEG-Interferon alfa-2a (Experimental)
  Interventions: Drug: Daclatasvir; Drug: Ribavirin; Drug: PEG-Interferon alfa 2a

INTERVENTIONS:
Drug: Daclatasvir — Tablets; oral; 30, 60, or 90 mg; once daily; up to 24 weeks
  Other Names: BMS-790052
Drug: Ribavirin — Tablets; oral; for patients weighing <75 kg, the total dose is 1000 mg per day (2 200-mg tablets in the morning and 3 200-mg tablets in the evening); for patients weighing >75 kg, the total dose is 1200 mg per day (3 200-mg tablets in morning and 3 200-mg tablets in evening); twice daily with food; 24 or 48 weeks depending on response
  Other Names: Copegus®
Drug: PEG-Interferon alfa 2a — Syringe, subcutaneous injection, 180 μg, once weekly, 24 or 48 weeks depending on response
  Other Names: Pegasys®; Pegylated interferon

SUMMARY:
The purpose of this open label study is to evaluate the safety and efficacy of daclatasvir plus pegylated interferon-alfa 2a and ribavirin in untreated hepatitis C virus in patients coinfected with HIV

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Key Inclusion Criteria:

* Males and females, 18 to 70 years of age
* Hepatitis C virus (HCV) genotype 1a or 1b
* HCV-treatment naive
* HCV RNA >10,000 IU/mL at screening
* HIV-1 infection (approximately 250 patients receiving highly active antiretroviral therapy [HAART], up to 50 patients not receiving HAART)
* For patients receiving HAART, HIV RNA must be below <40 copies/mL at screening and must be <400 copies/ml for at least 6 months prior to screening

Key Exclusion Criteria:

* Patients receiving HAART who first initiated antiretroviral therapy within the last 6 months of Day 1
* Patients receiving HAART who have changed their antiretroviral regimen due to safety or efficacy associated to HIV treatment within the last 3 months prior to Day 1. However, if changes are required to a patient's HAART regimen to meet the requirements of the protocol, these changes are allowed at the screening visit. The patient should wait a minimum of 1 month prior to Day 1 after a repeat of HIV viral load has been confirmed, <40 copies/ mL
* Use of prohibited HAART regimens within 1 month of Day 1 and throughout the treatment period of the trial (patients receiving HAART who have changed their antiretroviral regimen to initiate any HCV treatment within 6 weeks prior to Day 1)
* Laboratory values:

  1. Neutrophil count <1500 cells/μL (<1200 cells/ μL for Blacks)
  2. Platelet count <90,000 cells/μL
  3. Hemoglobin ≤12 g/dL for females, hemoglobin ≤13 g/dL for males
  4. Total bilirubin ≥34 μmol/L (or ≥2 mg/dL) unless a patient has a documented history of Gilbert's disease or antiretroviral regimen contains atazanavir
  5. Alanine aminotransferase ≥5*upper limit of normal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2011-12; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (70):
- United States (23):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Scripps Clinic, La Jolla, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Desert Medical Group Inc., Palm Springs, California
  - Ucsd Antiviral Research Center, San Diego, California
  - San Francisco Gen Hosp, San Francisco, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - Va Connecticut Healthcare System, West Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University Of Miami School Of Medicine, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Johns Hopkins University, Lutherville, Maryland
  - Saint Michael'S Medical Center, Newark, New Jersey
  - Upper Delaware Valley Infectious Diseases, Pc, Monticello, New York
  - Icahn School Of Medicine At Mount Sinai, New York, New York
  - Weill Cornell Medical College, New York, New York
  - James J Peters Vamc, The Bronx, New York
  - University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Morehead Medical Plaza, Charlotte, North Carolina
  - Amelia Court Hiv Research Clinic, Dallas, Texas
  - Baylor College Of Medicine, Houston, Texas
  - Texas Liver Institute, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Argentina (4):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Ciudad de Buenos Aires, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Prov de Santa Fe, Santa Fe Province
- Australia (4):
  - Local Institution, Darlinghurst, New South Wales
  - Local Institution, Darlinghurst Nsw, New South Wales
  - Local Institution, Clayton, Victoria
  - Local Institution, Parkville, Victoria
- Belgium (2):
  - Local Institution, Antwerp
  - Local Institution, Brussels
- Brazil (3):
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, São Paulo, São Paulo
- Canada (6):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Ottawa, Ontario
  - Local Institution, Torono, Ontario
  - Local Institution, Montreal, Quebec
- France (4):
  - Local Institution, Marseille
  - Local Institution, Montpellier
  - Local Institution, Paris
  - Local Institution, Pessac
- Germany (5):
  - Local Institution, Berlin
  - Local Institution, Bonn
  - Local Institution, Frankfurt
  - Local Institution, Frankfurt am Main
  - Local Institution, Hamburg
- Italy (4):
  - Local Institution, Brescia
  - Local Institution, Milan
  - Local Institution, Modena
  - Local Institution, Torino
- Puerto Rico (2):
  - Fundacion De Investigacion De Diego, San Juan
  - University Of Puerto Rico School Of Medicine, San Juan
- Russia (7):
  - Local Institution, Kaluga
  - Local Institution, Lipetsk
  - Local Institution, Moscow
  - Local Institution, Nizhny Novgorod
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov
  - Local Institution, Volgograd
- Spain (5):
  - Local Institution, Badalona, Barcelona
  - Local Institution, Barcelona
  - Local Institution, Córdoba
  - Local Institution, Madrid
  - Local Institution, Seville
- Local Institution, London, Greater London, United Kingdom

REFERENCES:
- [Derived] Sulkowski MS, Fessel WJ, Lazzarin A, Berenguer J, Zakharova N, Cheinquer H, Cote P, Dieterich D, Gadano A, Matthews G, Molina JM, Moreno C, Pineda JA, Pulido F, Rivero A, Rockstroh J, Hernandez D, McPhee F, Eley T, Liu Z, Mendez P, Hughes E, Noviello S, Ackerman P. Efficacy and safety of daclatasvir plus pegylated-interferon alfa 2a and ribavirin in previously untreated HCV subjects coinfected with HIV and HCV genotype-1: a Phase III, open-label study. Hepatol Int. 2017 Mar;11(2):188-198. doi: 10.1007/s12072-017-9788-z. Epub 2017 Feb 16. PMID 28210927
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 84 sites in 13 countries.
Pre-assignment Details: Of 549 participants enrolled, 301 were randomized to receive treatment. Of the 248 participants who were not randomized, 204 no longer met study criteria, and 44 discontinued due to other reasons.
Groups:
- Highly Active Anti-Retroviral Therapy (HAART):Daclatasvir,30mg: Participants taking HIV ritonavir-boosted protease inhibitors received daclatasvir tablets, 30 mg, orally once daily; peg-interferon alfa-2a (pegIFNalfa-2a) solution for injection, 180 µg, subcutaneously once weekly; and ribavirin tablets, orally twice daily with a total dose of 1000 mg for participants weighing <75 kg and 1200 mg for those weighing ≥75 kg, for up to 24 weeks. Participants without virologic response at Weeks 4 and 12 continued to receive pegIFNalfa-2a and ribavirin for a total duration of 48 weeks.
- HAART: Daclatasvir, 60 mg: Participants taking other HAART, including rilpivirine, received daclatasvir tablets, 60 mg, orally once daily; pegIFNalfa-2a solution for injection, 180 µg, subcutaneously once weekly; and ribavirin tablets orally twice daily with a total dose of 1000 mg for participants weighing <75 kg and 1200 mg for those weighing ≥75 kg, for up to 24 weeks. Participants without virologic response at Weeks 4 and 12 continued to receive pegIFNalfa-2a and ribavirin for a total duration of 48 weeks.
- HAART: Daclatasvir, 30 mg + 60 mg: Participants taking non-nucleoside reverse transcriptase inhibitors, except rilpivirine, received 2 daclatasvir tablets (1x30 mg and 1x60 mg), orally once daily; pegIFNalfa-2a solution for injection, 180 µg, subcutaneously, once weekly; and ribavirin tablets, orally twice daily for a total dose of 1000 mg for participants weighing <75 kg and 1200 mg for those weighing ≥75 kg, for up to 24 weeks. Participants without virologic response at Weeks 4 and 12 continued to receive pegIFNalfa-2a and ribavirin for a total duration of 48 weeks.
- Non--HAART Therapy: Participants not receiving HAART received daclatasvir tablets, 60 mg, orally, once daily; pegIFNalfa-2a solution for injection, 180 µg, subcutaneously, once weekly; and ribavirin tablets, orally, twice daily with a total dose of 1000 mg for participants weighing <75 kg and 1200 mg for those weighing ≥75 kg, for up to 24 weeks. Participants without virologic response at weeks 4 and 12 continued to receive pegIFNalfa-2a and ribavirin for a total duration of 48 weeks.
Period: Treatment Period
Arm/Group | Highly Active Anti-Retroviral Therapy (HAART):Daclatasvir,30mg | HAART: Daclatasvir, 60 mg | HAART: Daclatasvir, 30 mg + 60 mg | Non--HAART Therapy
Started | 132 | 39 | 106 | 24
Completed | 101 | 29 | 82 | 21
Not Completed | 31 | 10 | 24 | 3
Not completed — Lack of Efficacy | 12 | 4 | 14 | 1
Not completed — Adverse Event | 7 | 3 | 6 | 1
Not completed — Withdrawal by Subject | 5 | 1 | 1 | 0
Not completed — Patient Requested Discontinue Study drug | 4 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 2 | 2 | 0
Not completed — Patient no Longer Meets Study Criteria | 1 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0
Period: Follow-up Period
Arm/Group | Highly Active Anti-Retroviral Therapy (HAART):Daclatasvir,30mg | HAART: Daclatasvir, 60 mg | HAART: Daclatasvir, 30 mg + 60 mg | Non--HAART Therapy
Started | 121 | 34 | 102 | 24
Completed | 114 | 32 | 95 | 21
Not Completed | 7 | 2 | 7 | 3
Not completed — Withdrawal by Subject | 3 | 0 | 3 | 1
Not completed — Lost to Follow-up | 4 | 1 | 3 | 2
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Follow-up no longer required | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study therapy.
Groups:
- HAART Therapy: Daclatasvir, 60 mg: Participants taking other HAART, including rilpivirine, received daclatasvir tablets, 60 mg, orally once daily; pegIFNalfa-2a solution for injection, 180 µg, subcutaneously once weekly; and ribavirin tablets orally twice daily with a total dose of 1000 mg for participants weighing <75 kg and 1200 mg for those weighing ≥75 kg, for up to 24 weeks. Participants without virologic response at Weeks 4 and 12 continued to receive pegIFNalfa-2a and ribavirin for a total duration of 48 weeks.
- Non-HAART Therapy: Daclatasvir, 60 mg: Participants not receiving HAART received daclatasvir tablets, 60 mg, orally, once daily; pegIFNalfa-2a solution for injection, 180 µg, subcutaneously, once weekly; and ribavirin tablets, orally, twice daily with a total dose of 1000 mg for participants weighing <75 kg and 1200 mg for those weighing ≥75 kg, for up to 24 weeks. Participants without virologic response at weeks 4 and 12 continued to receive pegIFNalfa-2a and ribavirin for a total duration of 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Highly Active Anti-Retroviral Therapy (HAART):Daclatasvir,30mg | HAART Therapy: Daclatasvir, 60 mg | HAART: Daclatasvir, 30 mg + 60 mg | Non-HAART Therapy: Daclatasvir, 60 mg | Total
Number analyzed (Participants) | 132 | 39 | 106 | 24 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (9.72) | 47.9 (9.03) | 46.5 (9.42) | 36 (9.02) | 46.1 (9.90)
Age, Customized [Number; unit: participants]
  Younger than 65 years | 125 | 39 | 104 | 24 | 292
  65 years and older | 7 | 0 | 2 | 0 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 7 | 27 | 11 | 72
  Male | 105 | 32 | 79 | 13 | 229

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response at Follow-up Week 12 (SVR12)
Description: SVR12 was defined as hepatitis C virus (HCV) values lower than the lower limit of quantitation, target detected or target not detected at follow-up Week 12. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory. HAART=highly active antiretroviral therapy. SVR12 was defined as hepatitis C virus (HCV) values lower than the lower limit of quantitation, target detected or target not detected at follow-up Week 12. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory. HAART=highly active antiretroviral therapy.
Time Frame: Follow-up Week 12
Population: The analysis was performed in all participants who received at least 1 dose of study therapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- HAART: Daclatasvir, 30 mg + 60 mg: Participants taking non-nucleoside reverse transcriptase inhibitors, except rilpivirine, received daclatasvir tablets, 90 mg, orally once daily; pegIFNalfa-2a solution for injection, 180 µg, subcutaneously, once weekly; and ribavirin tablets, orally twice daily for a total dose of 1000 mg for participants weighing <75 kg and 1200 mg for those weighing ≥75 kg, for up to 24 weeks. Participants without virologic response at Weeks 4 and 12 continued to receive pegIFNalfa-2a and ribavirin for a total duration of 48 weeks.
- HAART Therapy: Daclatasvir 30 or 60 or 90 mg: Participants with prior exposure to HAART therapy, received daclatasvir tablets , either 30, 60 or 90 mg, orally, once daily; pegIFNalfa-2a solution for injection, 180 µg, subcutaneously, once weekly; and ribavirin tablets, orally twice daily for a total dose of 1000 mg for Participants weighing <75 kg and 1200 mg for those weighing ≥75 kg, for up to 24 weeks. Participants without virologic response at Weeks 4 and 12 continued to receive pegIFNalfa-2a and ribavirin for a total duration of 48 weeks.
Arm/Group | Highly Active Anti-Retroviral Therapy (HAART):Daclatasvir,30mg | HAART Therapy: Daclatasvir, 60 mg | HAART: Daclatasvir, 30 mg + 60 mg | HAART Therapy: Daclatasvir 30 or 60 or 90 mg | Non-HAART Therapy: Daclatasvir, 60 mg
Number analyzed (Participants) | 132 | 39 | 106 | 277 | 24
Percentage of participants | 75 [67.6 to 82.4] | 71.8 [57.7 to 85.9] | 71.7 [63.1 to 80.3] | 73.3 [68.1 to 78.5] | 87.5 [74.3 to 100]

2. Secondary Outcome: Percentage of Participants Who Achieved Hepatitis C Virus (HCV) RNA Levels Lower Than The Lower Limit of Quantitation (LLOQ), Target Detected (TD) or Target Not Detected (TND)
Description: Participants who achieved HCV RNA levels lower than the LLOQ i.e., 25 IU/ml, TD or TND. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory. HAART=highly active antiretroviral therapy.
Time Frame: Week 1, 2, 4, 6, 8, 12 and at both Weeks 4 and 12; end of treatment; and follow-up Weeks 12 and 24
Population: The analysis was performed in all participants who received at least 1 dose of study therapy. On-treatment virologic response rates were not significantly different from one another among 30 mg, 60 mg, and 90 mg groups in the HAART cohort, thus these groups were combined as per pre-specified analysis plan.
Measure: Number; unit: Percentage of participants
Arm/Group | HAART Therapy: Daclatasvir 30 or 60 or 90 mg | Non-HAART Therapy: Daclatasvir, 60 mg
Number analyzed (Participants) | 277 | 24
Percentage of participants
  Week 1 | 39.7 | 41.7
  Week 2 | 71.5 | 91.7
  Week 4 | 82.7 | 95.8
  Week 6 | 84.1 | 87.5
  Week 8 | 84.1 | 95.8
  Week 12 | 85.2 | 91.7
  Weeks 4 and 12 | 78.7 | 91.7
  End of treatment | 84.8 | 95.8
  Follow-up Week 12 | 73.3 | 87.5
  Follow-up Week 24 | 70.4 | 83.3

3. Secondary Outcome: Percentage of Participants Who Achieved Hepatitis C Virus (HCV) RNA Levels Lower Than the Lower Limit of Quantitation (LLOQ), Target Not Detected (TND)
Description: Participants who achieved HCV RNA levels lower than the LLOQ, TND. HCV RNA levels were measured by the Roche COBAS® TaqMan® HCV Test version 2.0 from the central laboratory. HAART=highly active antiretroviral therapy.
Time Frame: Week 1, 2, 4, 6, 8, and 12 and at both Weeks 4 and 12; end of treatment; and follow-up Weeks 12 and 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | HAART Therapy: Daclatasvir 30 or 60 or 90 mg | Non-HAART Therapy: Daclatasvir, 60 mg
Number analyzed (Participants) | 277 | 24
Percentage of participants
  Week 1 | 9 | 16.7
  Week 2 | 33.9 | 50
  Week 4 | 64.3 | 91.7
  Week 6 | 74.4 | 87.5
  Week 8 | 78 | 95.8
  Week 12 | 81.2 | 91.7
  Weeks 4 and 12 | 61.4 | 87.5
  End of treatment | 84.8 | 95.8
  Follow-up Week 12 | 73.3 | 87.5
  Follow-up Week 24 | 70.4 | 83.3

4. Secondary Outcome: Percentage of Participants Who Received Highly Active Antiretroviral Therapy (HAART), Maintained HIV RNA <40 Copies/mL, and Experienced Confirmed HIV RNA ≥400 Copies/mL
Description: Participants who received HAART, maintained HIV RNA <40 copies/mL, and experienced confirmed HIV RNA ≥ 400 copies/mL were determined.
Time Frame: End of treatment (up to Week 48)
Population: The analysis was performed in all participants who received at least 1 dose of study therapy
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- HAART Therapy: Daclatasvir, 30mg + 60 mg: Participants taking non-nucleoside reverse transcriptase inhibitors, except rilpivirine, received 2 daclatasvir tablets (1x30 mg and 1x60 mg),, orally once daily; pegIFNalfa-2a solution for injection, 180 µg, subcutaneously, once weekly; and ribavirin tablets, orally twice daily for a total dose of 1000 mg for participants weighing <75 kg and 1200 mg for those weighing ≥75 kg, for up to 24 weeks. Participants without virologic response at Weeks 4 and 12 continued to receive pegIFNalfa-2a and ribavirin for a total duration of 48 weeks.
Arm/Group | Highly Active Anti-Retroviral Therapy (HAART):Daclatasvir,30mg | HAART Therapy: Daclatasvir, 60 mg | HAART Therapy: Daclatasvir, 30mg + 60 mg | HAART Therapy: Daclatasvir 30 or 60 or 90 mg
Number analyzed (Participants) | 132 | 39 | 106 | 277
Percentage of participants
  HIV RNA <40 copies/mL | 88.6 [83.2 to 94.1] | 89.7 [80.2 to 99.3] | 93.4 [88.7 to 98.1] | 90.6 [87.2 to 94.1]
  HIV RNA ≥400 copies/mL | 0.0 [0.0 to 0.0] | 2.6 [0.0 to 7.5] | 0.0 [0.0 to 0.0] | 0.4 [0.0 to 1.1]

5. Secondary Outcome: Percentage of Participants With Sustained Virologic Response (SVR12) by rs12979860 Single Nucleotide Polymorphism (SNP) in the IL28B Gene
Description: Percentages calculated as number of responders/number who received treatment.
Time Frame: Follow-up Week 12
Population: The analysis was performed in all participants who received at least 1 dose of study therapy. Here 'n' signifies number of participants evaluable at the specified time-point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- HAART Therapy: Daclatasvir, 30 mg + 60 mg: Participants taking non-nucleoside reverse transcriptase inhibitors, except rilpivirine, received 2 daclatasvir tablets (1x30 mg and 1x60 mg), orally once daily; pegIFNalfa-2a solution for injection, 180 µg, subcutaneously, once weekly; and ribavirin tablets, orally twice daily for a total dose of 1000 mg for participants weighing <75 kg and 1200 mg for those weighing ≥75 kg, for up to 24 weeks. Participants without virologic response at Weeks 4 and 12 continued to receive pegIFNalfa-2a and ribavirin for a total duration of 48 weeks.
- HAART Therapy: Daclatasvir 30, 60 or 90 mg: Participants with prior exposure to HAART therapy, received daclatasvir tablets , either 30, 60 or 90 mg, orally, once daily; pegIFNalfa-2a solution for injection, 180 µg, subcutaneously, once weekly; and ribavirin tablets, orally twice daily for a total dose of 1000 mg for Participants weighing <75 kg and 1200 mg for those weighing ≥75 kg, for up to 24 weeks. Participants without virologic response at Weeks 4 and 12 continued to receive pegIFNalfa-2a and ribavirin for a total duration of 48 weeks.
Arm/Group | Highly Active Anti-Retroviral Therapy (HAART):Daclatasvir,30mg | HAART Therapy: Daclatasvir, 60 mg | HAART Therapy: Daclatasvir, 30 mg + 60 mg | HAART Therapy: Daclatasvir 30, 60 or 90 mg | Non-HAART Therapy: Daclatasvir, 60 mg
Number analyzed (Participants) | 132 | 39 | 106 | 277 | 24
Percentage of participants
  CC Genotype (n=36, 14, 39, 89, 6) | 94.4 [87.0 to 100.0] | 92.9 [79.4 to 100.0] | 79.5 [66.8 to 92.2] | 87.6 [80.8 to 94.5] | 100.0 [100.0 to 100.0]
  CT Genotype (n=72, 22, 50,144, 15) | 66.7 [55.8 to 77.6] | 63.6 [43.5 to 83.7] | 70.0 [57.3 to 82.7] | 67.4 [59.7 to 75.0] | 93.3 [80.7 to 100.0]
  TT Genotype (n=22, 3, 12, 37, 2) | 68.2 [48.7 to 87.6] | 33.3 [0.0 to 86.7] | 58.3 [30.4 to 86.2] | 62.2 [46.5 to 77.8] | 50.0 [0.0 to 100.0]
  Not reported (n=2, 0, 5, 7, 1) | 100.0 [100.0 to 100.0] | 0.0 [0.0 to 0.0] | 60.0 [17.1 to 100.0] | 71.4 [38.0 to 100.0] | 0.0 [0.0 to 0.0]

6. Secondary Outcome: Number of Participants Who Died and With Serious Adverse Event (SAEs), Grade 3 to 4 Adverse Events (AEs), and AEs Leading to Discontinuation
Description: Adverse event was defined as any new unfavorable symptom, sign, or disease or worsening of a pre-existing condition that does not necessarily have a causal relationship with treatment. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity, or drug dependency/abuse; was life-threating, an important medical event, or a congenital anomaly/birth defect; or required prolonged hospitalization. HAART=highly active antiretroviral therapy.
Time Frame: From Day 1 to 7 days post last dose of study treatment (up to Week 48)
Population: The analysis was performed in all participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Highly Active Anti-Retroviral Therapy (HAART):Daclatasvir,30mg | HAART Therapy: Daclatasvir, 60 mg | HAART Therapy: Daclatasvir, 30 mg + 60 mg | HAART Therapy: Daclatasvir 30 or 60 or 90 mg | Non-HAART Therapy: Daclatasvir, 60 mg
Number analyzed (Participants) | 132 | 39 | 106 | 277 | 24
Participants
  Deaths | 0 | 1 | 0 | 2 | 0
  SAEs | 12 | 6 | 6 | 24 | 0
  Grade 3 to 4 AEs | 46 | 12 | 35 | 93 | 4
  AEs leading to discontinuation | 7 | 4 | 6 | 17 | 1

ADVERSE EVENTS:
Time Frame: From Day 1 to 7 days post last dose of study treatment (up to Week 48)
Description: On-treatment period
Arm/Group | Highly Active Anti-Retroviral Therapy (HAART):Daclatasvir,30mg | HAART Therapy: Daclatasvir, 60 mg | HAART: Daclatasvir, 30 mg + 60 mg | Non-HAART Therapy: Daclatasvir, 60 mg
Serious Adverse Events (participants affected / at risk) | 12/132 | 6/39 | 6/106 | 0/24
Other Adverse Events (participants affected / at risk) | 122/132 | 38/39 | 100/106 | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Highly Active Anti-Retroviral Therapy (HAART):Daclatasvir,30mg (N=132) | HAART Therapy: Daclatasvir, 60 mg (N=39) | HAART: Daclatasvir, 30 mg + 60 mg (N=106) | Non-HAART Therapy: Daclatasvir, 60 mg (N=24)
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 0 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Laryngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 1 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Thrombophlebitis septic (Infections and infestations) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Highly Active Anti-Retroviral Therapy (HAART):Daclatasvir,30mg (N=132) | HAART Therapy: Daclatasvir, 60 mg (N=39) | HAART: Daclatasvir, 30 mg + 60 mg (N=106) | Non-HAART Therapy: Daclatasvir, 60 mg (N=24)
Abnormal dreams (Psychiatric disorders) | 1 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 19 | 4 | 8 | 5
Anxiety (Psychiatric disorders) | 5 | 3 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 20 | 3 | 14 | 4
Fatigue (General disorders) | 45 | 16 | 47 | 6
Genital herpes (Infections and infestations) | 1 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 36 | 10 | 17 | 3
Irritability (Psychiatric disorders) | 16 | 3 | 14 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 2 | 0
Chills (General disorders) | 5 | 4 | 6 | 1
Constipation (Gastrointestinal disorders) | 6 | 4 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 4 | 8 | 5
Diarrhoea (Gastrointestinal disorders) | 19 | 6 | 18 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 7 | 1
Nausea (Gastrointestinal disorders) | 24 | 10 | 21 | 4
Decreased appetite (Metabolism and nutrition disorders) | 32 | 9 | 27 | 5
Depression (Psychiatric disorders) | 20 | 5 | 17 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 3
Jaundice (Hepatobiliary disorders) | 7 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 4 | 2 | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 20 | 4 | 10 | 5
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 0
Sleep disorder (Psychiatric disorders) | 4 | 1 | 2 | 3
Asthenia (General disorders) | 40 | 7 | 19 | 12
Bronchitis (Infections and infestations) | 4 | 4 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 2 | 3 | 2 | 1
Depressed mood (Psychiatric disorders) | 3 | 2 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 42 | 7 | 35 | 4
Sciatica (Nervous system disorders) | 0 | 2 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 11 | 1 | 9 | 0
Dysgeusia (Nervous system disorders) | 9 | 4 | 7 | 0
Headache (Nervous system disorders) | 29 | 13 | 28 | 7
Hypertension (Vascular disorders) | 3 | 2 | 4 | 0
Influenza like illness (General disorders) | 28 | 14 | 15 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 26 | 5 | 14 | 5
Abdominal pain upper (Gastrointestinal disorders) | 8 | 0 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 2 | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 2 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 2 | 6 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 8 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 8 | 0 | 3 | 0
Pain (General disorders) | 6 | 3 | 4 | 0
Pharyngitis (Infections and infestations) | 3 | 2 | 1 | 0
Pyrexia (General disorders) | 28 | 6 | 19 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 1 | 8 | 0
Dry eye (Eye disorders) | 3 | 2 | 2 | 1
Lymphopenia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 3 | 14 | 6
Respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 2
Weight decreased (Investigations) | 14 | 3 | 8 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 32 | 10 | 34 | 4
Chest pain (General disorders) | 0 | 2 | 2 | 0
Dizziness (Nervous system disorders) | 11 | 3 | 7 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 3 | 0
Hyperthermia (General disorders) | 0 | 0 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 8 | 3 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 2
Vomiting (Gastrointestinal disorders) | 12 | 5 | 9 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.